CLINICAL TRIAL: NCT04373954
Title: Proposing Forgiveness Therapy for Those in Prison: An Intervention for Reducing Anger and Promoting Psychological Health
Brief Title: Proposing Forgiveness Therapy Within Prison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Department of Corrections, State of Wisconsin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0132; A173000 (Other: University of Wisconsin, Madison); EDUC/EDUC PSYCH (Other: University of Wisconsin, Madison)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Forgiveness
Keywords: Forgiveness

STUDY DESIGN:
Intervention Model Description: It is a cross-over design. For the first period of treatment, after the pretest, the experimental group received 6-month Forgiveness Therapy and the control group received 6-month alternative treatment-Carey Guides. The Carey Guides is a primary educational program deliberately picked by the Department of Corrections in Wisconsin. Some aspects emphasized in it include anti-social thinking, emotional regulation, moral reasoning, and so on. For the second period of treatment, after the post-test, the control group turned to the second experimental group and received 6-month Forgiveness Therapy, while the first experimental group had a rest for 6-month and then they finished the follow-up test or second post-test. For both experimental group and control group, they met once per week, one hour in a group setting. The remaining participants will be remeasured 12 months after the second period of treatment for one-year follow-up test.
Who Masked: Participant
Masking Description: Participants were randomly assigned to two treatments (Forgiveness Therapy and Carey Guides), without being informed about which type of treatment they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forgiveness Therapy (Experimental): 6-month Forgiveness Therapy; Participants meet once per week, in group setting.
  Interventions: Other: Forgiveness Therapy
- Carey Guides (Active Comparator): 6-month Carey Guides; Participants meet once per week, in group setting.
  Interventions: Other: Forgiveness Therapy; Other: Carey Guides

INTERVENTIONS:
Other: Forgiveness Therapy — The Forgiveness Therapy model mainly includes four stages: uncovering, decision, work and deepening. The book 8 Keys to Forgiveness (2015, a forgiveness therapy manual authored by Dr. Enright) is the basis for the therapy as a way to ensure that the treatment is uniformly founded on the forgiveness process developed at the University of Wisconsin-Madison.
Other: Carey Guides — The Carey Guides is a primary educational program deliberately chosen and approved by the Department of Corrections in Wisconsin, in which all inmates are encouraged (not required) to complete as they work toward custody reduction. Some aspects emphasized in it include anti-social thinking, emotional regulation, moral reasoning, and so on. It is the basis for the control group therapy as a way to ensure that the treatment has a uniform process as it is taught in the Department of Corrections (DOC) prison system.
  Arms: Carey Guides

SUMMARY:
Previous studies found that a large number of prisoners experienced unjust treatment from others, which can lead to deep inner pain or anger, prior to criminal perpetration. Such unresolved anger can deepen and linger, be turning to resentment (excessive anger) or rage (very intense, potentially violent anger), compromising one's psychological health and behavior and even contributing to their choice of crime. However, Forgiveness Therapy, as an empirically-verified treatment, can help reduce and even eliminate the excessive anger. Its positive effects have been scientifically supported by numerous studies within diverse populations. Therefore, in the prison context, similarly, the investigator hypothesizes that Forgiveness Therapy will lower rates of anger, depression, and anxiety and raise the levels of forgiveness, empathy, hope, and self-esteem for the experimental (Forgiveness Therapy) group as compared to the alternative treatment control group. This is based upon numerous studies that demonstrate the efficacy of Forgiveness Therapy with comparisons to other treatment methods. Further, the study team expects behavioral change by the men within the correctional institution, as measured by officers' observations as well as the number of misconducts in conduct reports on each participant and the time spent in restrictive housing.

This study is the second part of a two-tiered research project to propose a novel approach--Forgiveness Therapy--to corrections and aims to demonstrate the effectiveness of Forgiveness Therapy in reducing resentment and other negative psychological symptoms such as excessive anger, anxiety, and depression for the prison inmates.

A random sample of 24 participants, who have not participated in forgiveness workshops or forgiveness therapy, were taken from the Study 1(the investigator's previous research from the maximum-security prison of Columbia Correctional Institution "Examining Prison Inmates' Attitudes and Internal Emotional States"). These participants became 12 matched pairs (matched by the type of abuse, the severity of the abuse, and age at which the injustice occurred) with each member of the matched pair randomly assigned to the experimental group or control group. Each inmate participated voluntarily in this study.

Since this study is a continuation of Study 1, the investigator named this study as Study 2.

ELIGIBILITY:
Inclusion Criteria:

* Participants who enrolled in Study 1 and need to satisfy the criteria of:

  1. most serious stories of abuse against them; 2. the least forgiving; and 3. the most psychologically compromised. 4. Also, given the duration of psychological treatments, participants' release date will also be considered.

Exclusion Criteria:

* Inmates who have received Forgiveness Therapy before.
* Inmates would be released or transferred to other institutions during the 12-month treatment.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Anger | Baseline, 6 months, 12 months, 24 months
  National Institutes of Health PROMIS Measures of Anger (five items) was used. Items are statements about the frequency of feeling angry in the past seven days. An example is "In the past 7 days, I felt like I was ready to explode." Participants need to respond to each item on a 5-point scale from "Never" to "Always." The total scores for the anger scale range from 5 to 25. The higher scores a participant rated in one scale, the angrier participant was, in contrast with those who scored lower.
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Anxiety | Baseline, 6 months, 12 months, 24 months
  National Institutes of Health PROMIS Measures of Anxiety (seven items) was used. Items are statements about the frequency of feeling anxious in the past seven days. An example is "In the past seven days, I found it hard to focus on anything other than my anxiety." Participants need to respond to each item on a 5-point scale from "Never" to "Always." The total scores for the anxiety scale range from 5 to 35. The higher scores a participant rated in one scale, the more anxious participant was, in contrast with those who scored lower.
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Measures of Depression | Baseline, 6 months, 12 months, 24 months
  National Institutes of Health PROMIS Measures of Depression (eight items) was used. Items are statements about the frequency of feeling depressed in the past seven days. An example is "In the past seven days, I felt like a failure." Participants need to respond to each item on a 5-point scale from "Never" to "Always." The total scores for the anxiety scale range from 5 to 40. The higher scores a participant rated in one scale, the more depressed participant was, in contrast with those who scored lower.
Change in Score on Herth Hope Index | Baseline, 6 months, 12 months, 24 months
  The Herth Hope Index was used as an instrument. It has 12 items and assesses optimism toward the future with questions, such as "I have a positive outlook on life"; "I believe that each day has potential". These questions assess connectedness to positive expectations for the future, inter-connectedness with other people, and inner positive expectancy. Participants responded on a 4-point scale ranging from "strongly disagree" to "strongly agree." Two items need to be reversely coded, and the total hope score ranges from 12 to 48. A higher score means more hopefulness toward the future.
Change in Score on Enright Forgiveness Inventory | Baseline, 6 months, 12 months, 24 months
  Enright Forgiveness Inventory Short Form (30 items) was used as a measurement of forgiveness. It includes three subscales: affect, behavior, and cognition, with 10 items in each subscale. The introductory material at the beginning asks participants to focus on the worst injustice they experienced before their first imprisonment, and to indicate the person who unfairly treated them, time to event, degree of hurt and a brief description of the experience. Then participants were asked to think about the person who hurt them and rate the 30 items on a 6-point Likert scale ranging from "strongly disagree" to "strongly agree." Half of the items are negative statements, and reverse coding is done in the data analysis. An example of the positive items is "I feel warm toward him/her," and a negative one is "Regarding this person, I disapprove of him/her." The total forgiveness scores range from 30 to 180, with each subscale scores in the range of 10 to 60. A higher score means more forgiving.
Change in Score on Coopersmith Self-Esteem Inventory | Baseline, 6 months, 12 months, 24 months
  The Coopersmith Self-Esteem Inventory Form B (Adult Version), consisting of 25 true-false statements evaluating attitudes toward the self in the following domains: general self, social self, self and peers, self and parents, such as "I can make up my mind without too much trouble"; "I have a low opinion of myself". Whereas the original inventory was developed for use with children, Form B has been successfully modified and applied for adults both in college and industry. A participant gets 1 point for each "True" response and 0 point for each "False" response to 8 positive self-esteem statements, and the reverse points to 17 negative statements. Scores range from 0 to 25. A higher score means a higher self-esteem a participant has.
Change in Toronto Empathy Questionnaire Score | Baseline, 6 months, 12 months, 24 months
  The Toronto Empathy Questionnaire (TEQ) developed in partnership with the University of Toronto contains 16 items that cover both positive and absent responses of emotional empathy, such as "It upsets me to see someone being treated disrespectfully." "I enjoy making other people feel better." Participants responded on a 5-point scale ranging from "never" to "always." Half of the items need to be reversely coded, and the total empathy score ranges from 16 to 90. A higher score means a higher level of empathy.
Change in Score on Marlowe-Crowne Social Desirability Scale | Baseline, 6 months, 12 months, 24 months
  The Marlowe-Crowne Social Desirability Scale (20-item short version) was used here to measure if a participant is "faking good" to meet the social desirability in psychological tests. It also assesses the degree to which each participant is taking this set of questionnaires seriously or not. This 20-item short version of the Marlowe-Crowne Social Desirability Scale was developed by Strahan and Gerbasi, with 20 statements using a true/false response format. An example is "I never hesitate to go out of my way to help someone in trouble." A participant gets 1 point for each "True" response and 0 point for each "False" response to 10 socially desired statements, and the reverse points to 10 not socially desired statements. Scores range from 0 to 20. A higher score represents a higher tendency of "faking good" in the test.
Score on Maltreatment and Abuse Chronology of Exposure (MACE) Scale | Baseline
  The MACE scale includes 52 items and measures retrospectively ten types of maltreatment during each year of childhood from 1 to 18 years old. The ten subscales or types of maltreatment measured include: emotional neglect, non-verbal emotional abuse, parental physical maltreatment, parental verbal abuse, peer emotional abuse, peer physical bullying, physical neglect, sexual abuse, witnessing interparental violence, and witnessing violence to siblings.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enright, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Columbia Correctional Institution, Portage, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erzar T, Yu L, Enright RD, Kompan Erzar K. Childhood Victimization, Recent Injustice, Anger, and Forgiveness in a Sample of Imprisoned Male Offenders. Int J Offender Ther Comp Criminol. 2019 Jan;63(1):18-31. doi: 10.1177/0306624X18781782. Epub 2018 Jun 21. PMID 29926759
- [Background] Lee YR, Enright RD. A Forgiveness Intervention for Women With Fibromyalgia Who Were Abused in Childhood: A Pilot Study. Spiritual Clin Pract (Wash D C ). 2014 Sep;1(3):203-217. doi: 10.1037/scp0000025. Epub 2014 Aug 25. PMID 25914886
- [Background] Waltman MA, Russell DC, Coyle CT, Enright RD, Holter AC, M Swoboda C. The effects of a forgiveness intervention on patients with coronary artery disease. Psychol Health. 2009 Jan;24(1):11-27. doi: 10.1080/08870440903126371. PMID 20186637
- [Background] Hansen MJ, Enright RD, Baskin TW, Klatt J. A palliative care intervention in forgiveness therapy for elderly terminally ill cancer patients. J Palliat Care. 2009 Spring;25(1):51-60. PMID 19445342
- [Background] Reed GL, Enright RD. The effects of forgiveness therapy on depression, anxiety, and posttraumatic stress for women after spousal emotional abuse. J Consult Clin Psychol. 2006 Oct;74(5):920-9. doi: 10.1037/0022-006X.74.5.920. PMID 17032096
- [Background] Lin WF, Mack D, Enright RD, Krahn D, Baskin TW. Effects of forgiveness therapy on anger, mood, and vulnerability to substance use among inpatient substance-dependent clients. J Consult Clin Psychol. 2004 Dec;72(6):1114-21. doi: 10.1037/0022-006X.72.6.1114. PMID 15612857
- [Background] McKay KM, Hill MS, Freedman SR, Enright RD. Towards a feminist empowerment model of forgiveness psychotherapy. Psychotherapy (Chic). 2007 Mar;44(1):14-29. doi: 10.1037/0033-3204.44.1.14. PMID 22122165
- [Background] Enright, R. D., Erzar, T., Gambaro, M., Komoski, M. C., O'Boyle, J., Reed, G., & ... Yu, L. (2016). Proposing Forgiveness Therapy for those in Prison: An Intervention Strategy for Reducing Anger and Promoting Psychological Health. Journal of Forensic Psychology, 1, 116. DOI: 10.4172/2475-319X.1000116.
- [Background] Yu, L., Gambaro, M., Komoski, M. C., Song, M. J., Song, M., Teslik, M., Wollner, B., & Enright, R. D. (2018). The Silent Injustices against Men in Maximum Security Prison and the Need for Forgiveness Therapy: Two Case Studies. Journal of Forensic Psychology, 3, 137. DOI: 10.4172/2475-319X.1000137.
- See also: Project descriptions on this study — https://www.researchgate.net/project/Proposing-Forgiveness-Therapy-for-Those-in-Prison-An-Intervention-for-Reducing-Anger-and-Promoting-Psychological-Health